CLINICAL TRIAL: NCT03984682
Title: Impact of Joint Crisis Plan on the Duration of Isolation Measures in Psychiatry.
Brief Title: Impact of Joint Crisis Plan
Acronym: PLANCO-ISO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18PH221; ANSM (Other: 2019-A00062-55)
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Mental Disorders
Keywords: Joint Crisis Plan; Internalized Stigma of Mental Illness (ISMI); Isolation; physical restraint; Psychiatry
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients will benefit from regular care + Joint Crisis Plan
  Interventions: Procedure: Joint Crisis Plan
- Control group (No Intervention): Patients will benefit from regular care

INTERVENTIONS:
Procedure: Joint Crisis Plan — A Joint Crisis Plan will be drafted with the patient and a nurse
  Arms: Experimental group

SUMMARY:
For some patients in department psychiatric, isolation measures are put in place. But the measures is not pleasant for the patient or for the care team.

That's why care team are trying to find ways to improve patient care, including asking them how they would like to be treated.

One of the solutions is called the Joint Crisis Plan. A Joint Crisis Plan is a personalized procedure for a patient. It describes the attitude, the care, the measures in case of crisis with the patient and his family. Patients indicate their wishes regarding their care. However, there is no real scientific proof of the effectiveness of this Joint Crisis Plan, especially to reduce isolation measures.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate efficacy of the Joint Crisis Plan.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years
* Patients having had at least one isolation, restraint or forced hospitalization measure in the 24 months before inclusion
* Followed by nurses of a mobile team of psychiatry sector Saint Etienne
* Social security affiliation
* Signed informed consent

Exclusion Criteria:

* Patient having already had a Joint Crisis Plan for less than 6 months.
* Patient does not speak French
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Duration of isolation | Months: 12
  Measured in hours.

SECONDARY OUTCOMES:
Perception of constraint | Months: 12
  Measured by the MacArthur Coercion Scale. Each "True" = 0, and each "False" = 1, perceived cohesion scale score is between 0 and 5, Negative pressures scale score is between 0 and 6, Voice scale score is between 0 and 3, Affective Reactions to Hospitalization score is between 0 and 6.
Number of hospitalizations | Months: 12
Number of isolation | Months: 12
Number of physical restraints | Months: 12
Duration of physical restraint | Months: 12
  Measured in hours
Experience of discrimination and stigmatization | Months: 12
  Measured by the Internalized Stigma of Mental Illness. This scale is a 29 items scale with stigma graded on a 4 point scale (Strongly disagree-1, Disagree-2, Agree-3 and strongly agree-4) which are divided into fivecomponents/domains (alienation, stereotype endorsement, perceived discrimination, social withdrawal and stigma resistance). Higher scores indicate higher level of self stigma.
Number of violent events | Months: 12
Number of emergency room visits for psychiatric opinion | Months: 12
Adhesion and feeling of nurses in relation to Joint Crisis Plan | Months: 12
  Measured by focus-groups and individual interviews of nurses

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne QUENUM, Coordinating nurse, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No